CLINICAL TRIAL: NCT01455246
Title: Daptomycin + Meropenem Versus Ceftazidime in the Treatment of Nosocomial Spontaneous Bacterial Peritonitis: an Open, Randomized, Controlled Clinical Trial
Brief Title: Daptomycin + Meropenem Versus Ceftazidime in the Treatment of Nosocomial Spontaneous Bacterial Peritonitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decision of independent monitoring committee after interim analysis: Risk of failure significantly higher in ceftazidime group.
Sponsor: University of Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2059P; 2010-019625-34 (EudraCT Number)
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Cirrhosis; Ascites; Nosocomial Spontaneous Bacterial Peritonitis
Keywords: Cirrhosis; Nosocomial Spontaneous Bacterial Peritonitis; Ascites; Daptomycin; Meropenem; Ceftazidime; Nosocomial infection; Multi drug resistant bacteria; Sepsis; Albumin
MeSH Terms: conditions — Fibrosis; Ascites; Cross Infection; Sepsis | interventions — Daptomycin; Meropenem; Ceftazidime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daptomycin + Meropenem (Experimental): 30 patients with cirrhosis and nosocomial SBP
  Interventions: Drug: Daptomycin + Meropenem
- Ceftazidime (Active Comparator): 30 patients with cirrhosis and nosocomial SBP
  Interventions: Drug: Ceftazidime

INTERVENTIONS:
Drug: Daptomycin + Meropenem — Daptomycin will be administered at the dose of 6 mg/kg every 24 hours and 6 mg/kg every 48 hours for an estimated creatinine clearance (CKD-EPI) of > 30 ml/min and < 30 ml/min respectively. Meropenem will be administered at the dose of 1 g t.i.d., 1 g b.i.d., 0.5 g every 24 hours for an estimated creatinine clearance of >50 ml/min, 10-50 ml/min, and < 10 ml/min respectively. The treatment will go on for 7 days. In the patients without response to treatment after 48 hours will be added a rescue therapy with fluconazole. In patients in which cultures shown a bacterial species resistant to therapy, daptomycin and meropenem will be discontinued and replaced by a therapy based on antibiotic susceptibility of isolated species.
  Arms: Daptomycin + Meropenem
Drug: Ceftazidime — Ceftazidime will be administered at the dose of 2 g t.i.d, 2 g b.i.d and 2 g at every 24 hours by intravenous infusion for an estimated creatinine clearance (CKD-EPI) of >50 ml/min, 10-50 ml/min, and < 10 ml/min respectively. The treatment will go on for 7 days. In the patients without response to treatment after 48 hours, or in which cultures shown a bacterial species resistant to therapy, ceftazidime will be discontinued and replaced by a rescue therapy with meropenem and daptomycin as provided for the experimental arm
  Arms: Ceftazidime

SUMMARY:
Nosocomial spontaneous bacterial peritonitis (SBP) is frequently caused by multi drug resistant bacteria. Standard treatment of SBP could be ineffective. The aim of the study is to compare daptomycin + meropenem vs ceftazidime in the treatment of nosocomial SBP.

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP) is a well known complication in patients with liver cirrhosis and ascites. Nosocomial SBP is defined as SBP that occurs after 48 hours of hospitalization. It has been shown that patients with nosocomial SBP have a worse prognosis than patients with community-acquired SBP. It has also been shown that nosocomial SBP is frequently caused by multi drug resistant bacteria such as extended-spectrum-beta-lactamase (ESBL) producing enterobacteria or meticillin - resistant staphylococcus aureus. Currently the empirical treatment of SBP is the use of third generation cephalosporins or amoxicillin/clavulanic acid. In patients affected by nosocomial SBP these treatment could be ineffective. Up to now an empirical approach with a broader spectrum strategy (such as an association between meropenem and daptomycin) has never been compared to standard therapy in the treatment of nosocomial SBP. Thus, the aim of the study is to compare daptomycin + meropenem vs ceftazidime in the treatment of nosocomial SBP in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis and ascites
* Meets all criteria for nosocomial SBP as outlined below

  * Ascitic fluid polymorphonuclear cells count >250/mm3
  * Onset of signs and symptoms of infection after 72 hours of hospitalization

Exclusion Criteria:

* Hepatocellular carcinoma beyond the Milan criteria
* Abdominal surgery within 4 weeks
* Evidence of secondary peritonitis, pancreatitis or peritoneal carcinomatosis
* Significant heart or respiratory failure
* Allergy to ceftazidime, meropenem or daptomycin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary end-point of the study is the response to therapy | 48 hours and seven days
  The response to therapy is defined as the reduction of polymorphonuclear leukocytes (PMN) count in ascitic fluid more than 25 % from baseline after 48 hours and as a PMN count in ascitic fluid less then 250/mm³ after seven days.

SECONDARY OUTCOMES:
Mortality during hospitalization | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
30 days mortality | 30 days
90 days mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Angeli, MD, PhD, Principal Investigator — Dept. of Clinical and Experimenatl Medicine, University of Padova, Italy
Locations (1):
- Dept. of Clinical and Experimental Medicine, University of Padova, Padua, PD, Italy

REFERENCES:
- [Background] Rimola A, Garcia-Tsao G, Navasa M, Piddock LJ, Planas R, Bernard B, Inadomi JM. Diagnosis, treatment and prophylaxis of spontaneous bacterial peritonitis: a consensus document. International Ascites Club. J Hepatol. 2000 Jan;32(1):142-53. doi: 10.1016/s0168-8278(00)80201-9. No abstract available. PMID 10673079
- [Background] Fasolato S, Angeli P, Dallagnese L, Maresio G, Zola E, Mazza E, Salinas F, Dona S, Fagiuoli S, Sticca A, Zanus G, Cillo U, Frasson I, Destro C, Gatta A. Renal failure and bacterial infections in patients with cirrhosis: epidemiology and clinical features. Hepatology. 2007 Jan;45(1):223-9. doi: 10.1002/hep.21443. PMID 17187409
- [Background] Angeli P, Guarda S, Fasolato S, Miola E, Craighero R, Piccolo F, Antona C, Brollo L, Franchin M, Cillo U, Merkel C, Gatta A. Switch therapy with ciprofloxacin vs. intravenous ceftazidime in the treatment of spontaneous bacterial peritonitis in patients with cirrhosis: similar efficacy at lower cost. Aliment Pharmacol Ther. 2006 Jan 1;23(1):75-84. doi: 10.1111/j.1365-2036.2006.02706.x. PMID 16393283
- [Background] Cheong HS, Kang CI, Lee JA, Moon SY, Joung MK, Chung DR, Koh KC, Lee NY, Song JH, Peck KR. Clinical significance and outcome of nosocomial acquisition of spontaneous bacterial peritonitis in patients with liver cirrhosis. Clin Infect Dis. 2009 May 1;48(9):1230-6. doi: 10.1086/597585. PMID 19302016